CLINICAL TRIAL: NCT04223544
Title: Incidence of Influenza Infections and Determination of Vaccination Coverage Rate Among Hospital and GPs Healthcare Workers During the 2019/2020 Epidemic Season
Brief Title: Incidence of Influenza Infections and Determination of Vaccination Coverage Rate Among Healthcare Workers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Michał Jędrzejek, Principal Investigator, Wroclaw Medical University
Other Study IDs: 779/2019
Record Dates: First submitted 2020-01-06; First posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Influenza; Vaccination; Attitude of Health Personnel
Keywords: Influenza; Vaccination Coverage Rate; Healthcare Workers; General Practice; Point of Care Testing
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GPs Healthcare Workers
  Interventions: Diagnostic Test: Influenza POC and laboratory testing
- Hospital Healthcare Workers
  Interventions: Diagnostic Test: Influenza POC and laboratory testing

INTERVENTIONS:
Diagnostic Test: Influenza POC and laboratory testing — Participation in the study is voluntary and carried out after the consent of the examined person. The examination consists of: 1) completing the questionnaire and 2) taking the throat swab twice by the researcher. Two throat swab samples will be taken at the same time. Both samples will be used for virological examination to determine the presence of influenza virus material using non-invasive tests: one sample will be analyzed by a quick 'on-site' test - Flu SensDx kit, while the other sample will be transported to the laboratory, where the reverse transcriptase polymerase chain reaction (RT-PCR) - reference method - will be performed to confirm the presence of influenza genetic material. Swabs are planned to be collected during the 2019/2020 influenza epidemic season (January-March).

SUMMARY:
The main aim of research is to determine of the prevalence of influenza virus and influenza vaccination coverage rate among hospital and GPs healthcare workers.

Course of research:

Participation in the study is voluntary and carried out after the consent of the examined person. The examination consists of: 1) completing the questionnaire and 2) taking the throat swab twice by the researcher. Two throat swab samples will be taken at the same time. Both samples will be used for virological examination to determine the presence of influenza virus material using non-invasive tests: one sample will be analyzed by a quick 'on-site' test - Flu SensDx kit, while the other sample will be transported to the laboratory, where the reverse transcriptase polymerase chain reaction (RT-PCR) - reference method - will be performed to confirm the presence of influenza genetic material. Swabs are planned to be collected during the 2019/2020 influenza epidemic season (January-March).

In the last stage of the study, the results obtained from the survey questionnaire and the results of virological tests will be subject to statistical analysis and based on the data obtained, conclusions will be drawn from the study, indicating their practical application.

The results obtained from this study will be used to develop a quality improvement program to control influenza virus infection, which will improve the safety of both patients and medical staff.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare worker of selected General Practices or hospitals wards

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthcare workers of selected General Practices or hospitals wards: doctors, nurses, midwives
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-01-13 (Estimated); Primary Completion 2020-04-03 (Estimated); Study Completion 2020-04-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Influenza Infections | January-March 2020
  Incidence of influenza will be determined of results of POC and laboratory testing
Vaccination Coverage Rate | January-March 2020
  Vaccination Coverage Rate will be determined of survey questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Michal Jedrzejek, Principal Investigator — Family Medicine Department of Wroclaw Medical University
Locations (1):
- Family Medicine Department of Wroclaw Medical University, Wroclaw, Poland

REFERENCES:
- [Derived] Jedrzejek MJ, Mastalerz-Migas A, Janicka P. Incidence of Influenza Virus Infection among Wroclaw's Healthcare Workers in Pre-COVID-19 2019-2020 Influenza Season Using Novel Flu SensDx Device. Int J Environ Res Public Health. 2022 Mar 8;19(6):3159. doi: 10.3390/ijerph19063159. PMID 35328847